CLINICAL TRIAL: NCT02448381
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo Controlled Study to Determine the Efficacy of Topical SGX301 (Synthetic Hypericin) and Fluorescent Bulb-Light Irradiation for the Treatment of Cutaneous T-Cell Lymphoma
Brief Title: FLASH [Fluorescent Light Activated Synthetic Hypericin] Clinical Study: Topical SGX301 (Synthetic Hypericin) for the Treatment of Cutaneous T-Cell Lymphoma (Mycosis Fungoides)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPN-CTCL-01
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: CTCL; Mycosis fungoides; Hypericin; SGX301; MF
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — hypericin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SGX301 (Active Comparator): Three treatment cycles, each six (6) weeks followed by a two (2) week rest period. Treatment uses 0.25% SGX301 in USP Hydrophilic Ointment (or placebo) applied twice per week followed by fluorescent light therapy.
  Cycle 1: Patients randomized 2:1 to active/placebo will have three (3) index lesions treated and evaluated.
  Cycle 2: All patients will have three (3) index lesions treated and evaluated with active SGX301 ointment.
  Cycle 3: All patients will be given the opportunity to enter an open-label cycle of active SGX301 ointment treatment for all lesions (index and non-index).
  Interventions: Drug: SGX301 (synthetic hypericin)
- Placebo (Placebo Comparator): Placebo ointment is indistinguishable from ointment containing active SGX301 and is only used in Cycle 1. Treatment paradigm (ointment application and fluorescent light therapy) is identical.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGX301 (synthetic hypericin) — 0.25% SGX301 in USP Hydrophilic Ointment applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
  Other Names: Hypericin; Synthetic Hypericin
  Arms: SGX301
Drug: Placebo — USP Hydrophilic Ointment applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
  Arms: Placebo

SUMMARY:
To evaluate the use of SGX301, a topical photosensitizing agent, to treat patients with patch/plaque phase cutaneous T-cell lymphoma (mycosis fungoides).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of CTCL (mycosis fungoides), Stage IA, Stage IB, or Stage IIA.
* Subjects must have a minimum of three (3) evaluable, discrete lesions.
* Subjects must be willing to refrain from sunbathing for the duration of the study.

Exclusion Criteria:

* History of sun hypersensitivity and photosensitive dermatoses including porphyria, systemic lupus erythematosus, Sjögren's syndrome, xeroderma pigmentosum, polymorphous light eruptions or radiation therapy within 30 days of enrolling.
* Pregnancy or mothers who are breast feeding.
* Males and females not willing to use effective contraception.
* Unhealed sunburn.
* Subjects receiving topical steroids or other topical treatments for CTCL within 2 weeks.
* Subjects receiving systemic steroids, nitrogen mustard, psoralen UVA radiation therapy (PUVA), narrow band UVB light therapy (NB-UVB) or carmustine (BCNU) or other systemic therapies for CTCL within 3 weeks of enrollment.
* Subjects with significant history of systemic immunosuppression due to drugs or infection with HIV or HTLV 1.
* Subjects taking other investigational drugs or drugs of abuse within 30 days of entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - Therapeutics Clinical Research, San Diego, California
  - Olympian Clinical Research, Clearwater, Florida
  - Leon Medical Research, Miami, Florida
  - Medical Professional Clinical Research, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Tulane University, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rochester Skin Lymphoma Medical Group, Fairport, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - PMG Research of Wilmington, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Dermatology, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - INOVA Schar Cancer Institute, Fairfax, Virginia
  - Virginia Clinical Research, Norfolk, Virginia
  - Seattle Care Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Kim EJ, Mangold AR, DeSimone JA, Wong HK, Seminario-Vidal L, Guitart J, Appel J, Geskin L, Lain E, Korman NJ, Zeitouni N, Nikbakht N, Dawes K, Akilov O, Carter J, Shinohara M, Kuzel TM, Piette W, Bhatia N, Musiek A, Pariser D, Kim YH, Elston D, Boh E, Duvic M, Huen A, Pacheco T, Zwerner JP, Lee ST, Girardi M, Querfeld C, Bohjanen K, Olsen E, Wood GS, Rumage A, Donini O, Haulenbeek A, Schaber CJ, Straube R, Pullion C, Rook AH, Poligone B. Efficacy and Safety of Topical Hypericin Photodynamic Therapy for Early-Stage Cutaneous T-Cell Lymphoma (Mycosis Fungoides): The FLASH Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2022 Sep 1;158(9):1031-1039. doi: 10.1001/jamadermatol.2022.2749. PMID 35857290
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956
- See also: The National Organization for Rare Disorders — https://www.rarediseases.org/
- See also: The Cutaneous Lymphoma Foundation — http://www.clfoundation.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- SGX301: Three treatment cycles, each six (6) weeks followed by a two (2) week rest period. Treatment uses 0.25% SGX301 in USP Hydrophilic Ointment (or placebo) applied twice per week followed by fluorescent light therapy.
  Cycle 1: Patients randomized 2:1 to active/placebo will have three (3) index lesions treated and evaluated.
  Cycle 2: All patients will have three (3) index lesions treated and evaluated with active SGX301 ointment.
  Cycle 3: All patients will be given the opportunity to enter an open-label cycle of active SGX301 ointment treatment for all lesions (index and non-index).
  SGX301 (synthetic hypericin): 0.25% SGX301 in USP Hydrophilic Ointment applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
- Placebo: Placebo ointment is indistinguishable from ointment containing active SGX301 and is only used in Cycle 1. Treatment paradigm (ointment application and fluorescent light therapy) is identical.
  Placebo: USP Hydrophilic Ointment applied twice per week, covered by opaque bandage for 18-24 hours, then treated with an initial dose of 12 J/cm^2 fluorescent light.
Period: Overall Study
Arm/Group | SGX301 | Placebo
Started | 118 | 51
Randomized, Not Treated | 2 | 1
Cycle 1 | 116 | 50
Cycle 2 | 110 | 45
Cycle 3 | 78 | 32
Follow-up Period | 98 | 39
Completed | 83 | 32
Not Completed | 35 | 19
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 16 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Noncompliance with Study Procedures | 2 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was defined as all participants that were treated with at least one dose of treatment (SGX301 or Placebo)
Groups:
- Total: Total of all reporting groups
Arm/Group | SGX301 | Placebo | Total
Number analyzed (Participants) | 116 | 50 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (15.94) | 59.4 (16.26) | 58.4 (16.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 23 | 70
  Male | 69 | 27 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 3 | 13
  Not Hispanic or Latino | 103 | 45 | 148
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 84 | 36 | 120
  Black or African American | 27 | 12 | 39
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 0 | 2 | 2
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders and Non-Responders With a Treatment Response in 3 Treated Lesions as Defined as a ≥50% Improvement in the Composite Assessment of Index Lesion Disease Severity (CAILS) Score When Compared to Patients Receiving Placebo
Description: The percentage of patients achieving a treatment response in each of the 2 treatment groups. A treatment response was defined as a ≥50% improvement in CAILS score at Week 8 when compared to the CAILS score at baseline.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.
  The overall CAILS score was calculated by adding the total score as described above for each of the 3 lesions. The overall CAILS score has a range of 0 to 111. A lower score means a better outcome.
Time Frame: 8 weeks
Population: The analysis population was defined as all participants that were treated with at least one dose of treatment (SGX301 or Placebo)
Measure: Count of Participants; unit: Participants
Groups:
- SGX301: Three treatment cycles, each six (6) weeks followed by a two (2) week rest period. Treatment uses 0.25% SGX301 in USP Hydrophilic Ointment (or placebo) applied twice per week followed by fluorescent light therapy.
  Cycle 1: Patients have three (3) index lesions treated with SGX301 (0.25% synthetic hypericin in USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
- Placebo: Placebo ointment is indistinguishable from ointment containing active SGX301 and is only used in Cycle 1. Treatment paradigm (ointment application and fluorescent light therapy) is identical.
  Cycle 1: Patients have three (3) index lesions treated with Placebo (USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
Arm/Group | SGX301 | Placebo
Number analyzed (Participants) | 116 | 50
Participants
  Responder | 19 | 2
  Non-responder | 97 | 48
Statistical Analysis 1: Comparison: SGX301 vs Placebo; Test type: Superiority; p = 0.04, Regression, Logistic

2. Secondary Outcome: Number of Responders and Non-Responders With a Treatment Response in 3 Treated Lesions as Measured by the Composite Assessment of Index Lesion Disease Severity (CAILS) Score (Cycle 1 and 2 SGX301 vs Cycle 1 Placebo)
Description: The percentage of patients achieving a treatment response at Week 16 that received SGX301 for both Cycle 1 and 2 compared to the response rate in patients that received Placebo in Cycle 1.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score was measured as previously described.
Time Frame: 16 weeks
Population: The analysis population was defined as all participants that were treated with at least one dose of treatment (SGX301) in Cycle 2
Measure: Count of Participants; unit: Participants
Groups:
- SGX301 (Cycle 1 & 2 = SGX301): Three treatment cycles, each six (6) weeks followed by a two (2) week rest period. Treatment uses 0.25% SGX301 in USP Hydrophilic Ointment (or placebo) applied twice per week followed by fluorescent light therapy.
  Cycle 1: Patients have three (3) index lesions treated with SGX301 (0.25% synthetic hypericin in USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
  Cycle 2: Patients have three (3) index lesions treated with SGX301 (0.25% synthetic hypericin in USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
- Placebo (Cycle 1): Placebo ointment is indistinguishable from ointment containing active SGX301 and is only used in Cycle 1. Treatment paradigm (ointment application and fluorescent light therapy) is identical.
  Cycle 1: Patients have three (3) index lesions treated with Placebo (USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 12 J/cm^2 fluorescent light.
Arm/Group | SGX301 (Cycle 1 & 2 = SGX301) | Placebo (Cycle 1)
Number analyzed (Participants) | 110 | 50
Participants
  Responder | 44 | 2
  Non-responder | 66 | 48
Statistical Analysis 1: Comparison: SGX301 (Cycle 1 & 2 = SGX301) vs Placebo (Cycle 1); Test type: Superiority; p < 0.0001, Regression, Logistic

3. Secondary Outcome: Number of Responders and Non-Responders With a Treatment Response of 3 Treated Lesions as Measured by the Composite Assessment of Index Lesion Disease Severity (CAILS) Score in Patients Who Received 3 Cycles of SGX301
Description: The percentage of patients achieving a treatment response at Week 24 compared at Week 16 in SGX301 treatment group. A treatment response was defined as a ≥50% improvement in CAILS score when compared to the CAILS score at baseline.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score was measured as previously described.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- SGX301 (Cycle 1, 2 & 3 = SGX301): Three treatment cycles, each six (6) weeks followed by a two (2) week rest period. Treatment uses 0.25% SGX301 in USP Hydrophilic Ointment (or placebo) applied twice per week followed by fluorescent light therapy.
  Cycle 1: Patients have three (3) index lesions treated with SGX301 (0.25% synthetic hypericin in USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
  Cycle 2: Patients have three (3) index lesions treated with SGX301 (0.25% synthetic hypericin in USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
  Cycle 3: Patients have three (3) index lesions treated with SGX301 (0.25% synthetic hypericin in USP Hydrophilic Ointment) applied twice per week, covered by opaque bandage for 12-24 hours, then treated with an initial dose of 5 J/cm^2 fluorescent light.
Arm/Group | SGX301 (Cycle 1, 2 & 3 = SGX301)
Number analyzed (Participants) | 78
Participants
  Responder | 38
  Non-responder | 40
Statistical Analysis 1: Comparison: SGX301 (Cycle 1, 2 & 3 = SGX301); Test type: Superiority; p = 0.046, McNemar

4. Secondary Outcome: Patch Lesion Response Rates With Extended Treatment (Cycle 1 & 2 SGX301 vs Cycle 1 Placebo)
Description: The proportion of patch lesions achieving a treatment response at Week 16 in the SGX301 treatment group compared to Week 8 in the Placebo treatment group. A treatment response was defined as a ≥50% improvement in CAILS score when compared to the CAILS score at baseline for individual lesions.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score was measured as previously described.
Time Frame: 16 weeks
Population: as for outcome 2
Measure: Number; unit: lesions with response
Units Other Than Participants: lesions
Arm/Group | SGX301 (Cycle 1 & 2 = SGX301) | Placebo (Cycle 1)
Number analyzed (Participants) | 110 | 50
Number analyzed (lesions) | 178 | 85
lesions with response | 65 | 14
Statistical Analysis 1: Comparison: SGX301 (Cycle 1 & 2 = SGX301) vs Placebo (Cycle 1); Test type: Superiority; p = 0.0009, Fisher Exact

5. Secondary Outcome: Plaque Lesion Response Rates With Extended Treatment (Cycle 1 & 2 SGX301 vs Cycle 1 Placebo)
Description: The proportion of plaque lesions achieving a treatment response at Week 16 in the SGX301 treatment group compared to Week 8 in the Placebo treatment group. A treatment response was defined as a ≥50% improvement in CAILS score when compared to the CAILS score at baseline for individual lesions.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score was measured as previously described.
Time Frame: 16 weeks
Population: The analysis population was defined as all lesions that were treated with at least one dose of treatment (SGX301) in Cycle 2
Measure: Number; unit: lesions with response
Units Other Than Participants: lesions
Arm/Group | SGX301 (Cycle 1 & 2 = SGX301) | Placebo (Cycle 1)
Number analyzed (Participants) | 110 | 50
Number analyzed (lesions) | 152 | 65
lesions with response | 64 | 7
Statistical Analysis 1: Comparison: SGX301 (Cycle 1 & 2 = SGX301) vs Placebo (Cycle 1); Test type: Superiority; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (SGX301 or Placebo) until 1 month following the participant's last evaluation visit (Cycle 1 = 8 weeks, Cycle 2 = 16 weeks, Cycle 3 = 24 weeks)
Groups:
- Cycle 1 - SGX301: Patients treated with SGX301 in Cycle 1.
- Cycle 1 - Placebo: Patients treated with Placebo in Cycle 1. Cycle 1 is the only cycle that used Placebo.
- Cycle 2 - SGX301: Patients treated with SGX301 in Cycle 2. Since all patients received SGX301 in Cycle 2, this includes 45 patients that received Placebo in Cycle 1 and 110 patients that continued to receive SGX301 in Cycle 2.
- Cycle 3 - SGX301: Patients treated with SGX301 in Cycle 3. Since all patients received SGX301 in Cycle 3, this includes 32 patients that received Placebo in Cycle 1 and 78 patients that continued to receive SGX301 in Cycle 3.
- Overall SGX301: Any participant that received at least one dose of SGX301 during any cycle of the trial.
Arm/Group | Cycle 1 - SGX301 | Cycle 1 - Placebo | Cycle 2 - SGX301 | Cycle 3 - SGX301 | Overall SGX301
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/50 | 0/155 | 0/110 | 0/161
Serious Adverse Events (participants affected / at risk) | 1/116 | 1/50 | 0/155 | 3/110 | 4/161
Other Adverse Events (participants affected / at risk) | 56/116 | 26/50 | 66/155 | 49/110 | 108/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 - SGX301 (N=116) | Cycle 1 - Placebo (N=50) | Cycle 2 - SGX301 (N=155) | Cycle 3 - SGX301 (N=110) | Overall SGX301 (N=161)
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Gastritis alcoholic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 - SGX301 (N=116) | Cycle 1 - Placebo (N=50) | Cycle 2 - SGX301 (N=155) | Cycle 3 - SGX301 (N=110) | Overall SGX301 (N=161)
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2 | 2 | 5 | 12
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 1 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 4 | 2 | 2 | 12
Viral upper respiratory tract infection (Infections and infestations) | 4 | 0 | 4 | 4 | 11
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 3 | 7
Urinary tract infection (Infections and infestations) | 1 | 2 | 3 | 0 | 4
Influenza (Infections and infestations) | 0 | 2 | 1 | 2 | 3
Application site pain (General disorders) | 8 | 2 | 5 | 6 | 16
Application site pruritus (General disorders) | 5 | 1 | 5 | 0 | 9
Fatigue (General disorders) | 3 | 1 | 3 | 2 | 8
Application site paraesthesia (General disorders) | 6 | 0 | 2 | 2 | 7
Pain (General disorders) | 3 | 0 | 2 | 0 | 5
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 3 | 0 | 6
Headache (Nervous system disorders) | 5 | 3 | 5 | 2 | 10
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 2 | 6
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 5 | 5 | 17
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 | 2 | 4 | 5 | 14
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6 | 4 | 11
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 2 | 5
Eye disorders (Eye disorders) | 3 | 0 | 2 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT02448381/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT02448381/SAP_001.pdf